CLINICAL TRIAL: NCT06456671
Title: Examining the Generality of Laboratory-based Findings and Their Moderators Using Diverse Samples From the International Tobacco Control (ITC) Policy Evaluation Project Cohorts - Study 3a
Brief Title: Examining the Generality of Laboratory-based Findings and Their Moderators in the ITC Study
Acronym: MUSC-R 3a
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Medical University of South Carolina (Other); University of Waterloo (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Roberta Freitas-Lemos, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB #24-520; 5P01CA200512 (NIH)
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-08

CONDITIONS: Cigarette Smoking; Nicotine Vaping
MeSH Terms: conditions — Cigarette Smoking; Vaping

STUDY DESIGN:
Intervention Model Description: Participants will complete seven Experimental Tobacco Marketplace conditions. Conventional cigarette price will be parametrically increased, and the purchasing of alternative products measured. Alternative products (i.e. nicotine vaping products, heated tobacco products and nicotine pouches) will be available at different prices in separate conditions (i.e., ½ market price and market price).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exclusive cigarette smokers (Experimental): Exclusive cigarette smokers will be recruited and will be exposed to all of the conditions described in the intervention section.
  Interventions: Other: All nicotine/ tobacco products at market price; Other: Nicotine vaping products at 1/2 market price; Other: Heated tobacco products at 1/2 market price.; Other: Nicotine pouch products at 1/2 market price.
- Dual cigarette/ nicotine vaping product users (Experimental): Dual cigarette and nicotine vaping product users will be recruited and will be exposed to all of the conditions described in the intervention section.
  Interventions: Other: All nicotine/ tobacco products at market price; Other: Nicotine vaping products at 1/2 market price; Other: Heated tobacco products at 1/2 market price.; Other: Nicotine pouch products at 1/2 market price.

INTERVENTIONS:
Other: All nicotine/ tobacco products at market price — Nicotine/tobacco products available in the Experimental Tobacco Marketplace at market price. Note that all participants will complete all the specified conditions.
Other: Nicotine vaping products at 1/2 market price — Availability of nicotine vaping products in the Experimental Tobacco Marketplace at 1/2 market price. Other nicotine/tobacco products at market price. Note that all participants will complete all the specified conditions.
Other: Heated tobacco products at 1/2 market price. — Availability of heated tobacco products in the Experimental Tobacco Marketplace at 1/2 market price. Other nicotine/tobacco products at market price. Note that all participants will complete all the specified conditions.
Other: Nicotine pouch products at 1/2 market price. — Availability of heated tobacco products in the Experimental Tobacco Marketplace at 1/2 market price. Other nicotine/tobacco products at market price. Note that all participants will complete all the specified conditions.

SUMMARY:
This study will investigate the relative appeal (abuse liability) of novel tobacco products, how the appeal is modulated by relative price, user type, and how novel products may substitute for one another.

DETAILED DESCRIPTION:
An important aim of tobacco control is to reduce demand for the most harmful products. Therefore, a priori knowledge of substitutability across novel and widely used tobacco products may forecast the impact of policies on product switching. This study will use a novel method, the Experimental Tobacco Marketplace (ETM), to characterize the relative substitutability and appeal (abuse liability) of tobacco products (e.g., conventional cigarettes, nicotine vaping products [NVP], heated tobacco products [HTP], and nicotine pouch products [NPP]), and how the appeal is modulated by relative price, user type, and regulatory environment. Exclusive cigarette smokers and dual cigarette/NVP users, stratified by age, will complete multiple scenarios in the ETM.

ELIGIBILITY:
Inclusion Criteria:

* From CA, US, or EN
* At least 21 years old
* Smoking daily
* Smoking mostly or about equal amounts of factory-made cigarettes
* Does not currently vape (for exclusive smokers only)
* Vapes Daily (for dual users only)

Exclusion Criteria:

* There will be no additional exclusion criteria for this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Cigarette demand | 1 day
  Participants will complete purchasing trials in an Experimental Tobacco Marketplace (ETM) with cigarettes increasing in price. Other product prices in the ETM will depend on the experimental condition. The degree to which other nicotine/tobacco products substitute for conventional cigarettes as a function of novel product (e.g. nicotine vaping products, heated tobacco products, nicotine pouch products) prices will be assessed.
  To obtain dependent measures of demand, participants' purchasing of the price-manipulated commodity in the ETM task will be fit to a modified exponential equation to quantify the relationship between the price of each commodity and purchasing: Q=Q0*10k(exp(-αQ0C)-1) where Q is purchasing of the commodity, C is the price, Q0 is the derived initial purchasing without cost constraints (demand intensity), k is the span of the function in logarithmic units, and α is the demand elasticity.
Nicotine/tobacco products substitution | 1 day
  Participants will complete purchasing trials in an Experimental Tobacco Marketplace (ETM) with cigarettes increasing in price. Other product prices in the ETM will depend on the experimental condition. The degree to which other nicotine/tobacco products substitute for conventional cigarettes as a function of novel product (e.g. nicotine vaping products, heated tobacco products, nicotine pouch products) prices will be assessed.
  To obtain estimates of substitution of price-constant products in the different ETM conditions, the investigators will use ordinary least squares regression to model the relationship of the price-manipulated product to predict total quantity purchased of the price-constant product.

CONTACTS AND LOCATIONS:
Overall Officials: Warren K Bickel, Ph.D., Principal Investigator — Fralin Biomedical Research Institute at VTC
Locations (1):
- Fralin Biomedical Research Institute, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
The study team will share de-identified data upon request.